CLINICAL TRIAL: NCT02521922
Title: Feasibility Study for Automated Monitoring of Vital Signs Measurements in the In-Patient Hospital Setting
Brief Title: Vital Signs Patch Early Feasibility and Usability Study
Acronym: VSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeWatch Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VSP-F001v1.2
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Vital Signs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VSP Study Participants (Experimental): Vital Signs Patch system study participants. Each study participant will receive the VSP System - NEHB Configuration and then the VSP System - PAL Configuration. Vital signs will be taken and adhesive will be assessed for each participant for each configuration.
  Interventions: Device: VSP System - NEHB Configuration; Device: VSP System - PAL Configuration

INTERVENTIONS:
Device: VSP System - NEHB Configuration — VSP System - NEHB Configuration will take and record participant vital signs. NEHB is the last name of the physician who developed the configuration. It is not an acronym.
Device: VSP System - PAL Configuration — VSP System - PAL Configuration will take and record patient vital signs. PAL is the name created by the engineering team of this device. It is not an acronym.

SUMMARY:
To assess the feasibility and usability of the VSP System in the in-patient hospital setting to monitor vital signs using a patch, brain, gateway, and console. The VSP System will be incorporated into the study site's Information Technology infrastructure.

DETAILED DESCRIPTION:
The primary objective of this clinical feasibility study is to evaluate the feasibility of the Vital Signs Patch System (VSP). The VSP will be incorporated into the study site's Information Technology infrastructure and worn by in-patients for a minimum of 3 days and for the duration of their hospital stay up to 7 days.

The VSP will take and monitor vital signs in addition to the normal equipment the facility uses to monitor and take vital signs. This study will not be assessing safety and no comparator groups will be used. As this study will not be treating any particular disease or condition, no randomization or blinding is required. Subjects will be chosen as they are admitted in accordance with the general population characteristics, inclusion and exclusion criteria and willingness to sign the Informed Consent.

This clinical study involves a device with no additional drugs administered.

During this study, a single VSP System patch will be worn for up to 48 hours. The first patch will be placed using the NEHB configuration. After the first 48 hours, the NEHB-configured patch will be replaced with a new patch in the PAL configuration. The second patch can remain on the subject for the duration of the subject's hospital stay, or up to seven (7) consecutive days. Individual patient use will determine the duration of time that the second patch can be worn.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female in-patients with vital signs considered 'stable' by clinical caregivers.

Exclusion Criteria:

* Pediatric patients
* Female patients who are pregnant
* Patients with internal or external defibrillators
* Patients who have undergone surgery and still have a fresh incision on the chest.
* Patients with skin damage on the chest such as burns, irritation, infections, wounds, etc.
* Patients in the Critical Care Unit (CCU)
* Patients who otherwise satisfy any of the contraindications associated with the VSP system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04-16; Primary Completion 2016-06-09 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Composite Outcome Measure - 100% Successful Vital Signs Acquisition | Up to seven days
  Successful acquisition of Temperature, Heart Rate, ECG, Respiration, and SpO2 daily for the inpatient stay of the subject up to seven days. Success is achieved if all vital signs are obtained on a study participant. It is a composite result.

SECONDARY OUTCOMES:
Composite Outcome Measure - Adhesive Performance - Measurement of skin irritation resulting from adhesive used with electrodes. | Up to seven days
  Successful performance of the adhesive of the patch throughout the study for each subject. Subject skin will be checked daily to determine if irritation has resulted where the electrodes have been placed. The results will be either positive or negative for skin irritation. This is a composite outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, M.D., Principal Investigator — Mt. Sinai Medical Center; Marie Noelle-Langan, M.D., Principal Investigator — Mt. Sinai Medical Center
Locations (1):
- Mt. Sinai Medical Center, New York, New York, United States